CLINICAL TRIAL: NCT04732832
Title: Risk of Hepatitis C Virus Reinfection in Hemodialysis Patients With Chronic Hepatitis C Achieving Sustained Virologic Response Following Antiviral Therapy
Brief Title: HCV Reinfection in HD Patients Achieving SVR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202012090RINC
Record Dates: First submitted 2021-01-26; First posted 2021-02-01 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Hepatitis C Virus Infection; Hepatitis C Virus Infection, Response to Therapy of; Hemodialysis Complication
Keywords: Hepatitis C virus; Hemodialysis; Sustained virologic response; Reinfection
MeSH Terms: conditions — Hepatitis C; Reinfection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Among the hemodialysis units, the global incidence of HCV infection ranges from 1.2% to 2.9%. Data regarding the long-term risk of reinfection among hemodialysis patients achieving SVR are limited. To our best knowledge, only one study assessed the long-term negativity of serum HCV RNA in hemodialysis patients who achieved SVR after IFN-based therapies. With a median follow-up of 48 months following SVR, the life-time cumulative survival for HCV RNA negativity was 86% among the 121 participants who were on maintenance dialysis. Furthermore, the life-time cumulative survival for HCV RNA negativity was 95% among the 45 participants who underwent renal transplantation from HCV-negative donors. Because the literatures regarding the long-term follow-up of viral outcome, the patient numbers to be recruited are still limited, and all studies are focused on IFN-based treatment, we aim to assess the long-term risk of HCV reinfection in hemodialysis patients attaining SVR by IFN-based or IFN-free therapies.

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) infection is an important public health problem. Compared to the global prevalence of HCV infection to be around 1.0%, the prevalence of HCV infection in hemodialysis patients is around 10%. The high prevalence of HCV infection in hemodialysis patients receiving long-term renal replacement therapy may be reasoned by the nosocomial transmission in hemodialysis units. If chronic HCV infection is left untreated, the survival, hospitalization and the quality of life are significantly compromised in hemodialysis patients. In contrast, the survival is improved following successful treatment-induced HCV clearance Interferon (IFN)-based therapy is the treatment of choice for hemodialysis patients with HCV infection in earlier years. However, the treatment responses are far from ideal and the treatment-emergent adverse events (AEs) are frequently encountered, making the global treatment uptake rate by IFN-based therapies to be only 1.5%. Based on the excellent efficacy and safety, IFN-free direct acting antivirals (DAAs) have been the mainstay of therapy for HCV. Furthermore, the world health organization (WHO) has set the goal of global HCV elimination by 2030. The microelimination of HCV among hemodialysis patients is also listed as the prioritized target by WHO.

The updated definition of sustained virologic response (SVR) is the presence of serum undetectable HCV RNA level at week 12 after the stopping of antiviral therapy. However, the consensus in Taiwan mandates that hemodialysis patients who achieve SVR at off-therapy week 24 can be moved from HCV-segregated zone to cleat zone in hemodialysis unit, instead of the global definition of off-therapy week 12. The delay of bed-transfer from HCV-infective zone to clear zone might increase the risk of reinfection in hemodialysis patients achieving SVR. Therefore, we aim to assess the risk of short-term of HCV reinfection in hemodialysis patients achieving SVR at week 12 after antiviral therapy, which may be great relevance and importance for health policy making.

Among the hemodialysis units, the global incidence of HCV infection ranges from 1.2% to 2.9%. Data regarding the long-term risk of reinfection among hemodialysis patients achieving SVR are limited. To our best knowledge, only one study assessed the long-term negativity of serum HCV RNA in hemodialysis patients who achieved SVR after IFN-based therapies. With a median follow-up of 48 months following SVR, the life-time cumulative survival for HCV RNA negativity was 86% among the 121 participants who were on maintenance dialysis. Furthermore, the life-time cumulative survival for HCV RNA negativity was 95% among the 45 participants who underwent renal transplantation from HCV-negative donors. Because the literatures regarding the long-term follow-up of viral outcome, the patient numbers to be recruited are still limited, and all studies are focused on IFN-based treatment, we aim to assess the long-term risk of HCV reinfection in hemodialysis patients attaining SVR by IFN-based or IFN-free therapies.

ELIGIBILITY:
Inclusion Criteria:

* Age old than 20 years old
* Patients receiving hemodialysis during interferon (IFN)-based or IFN-free antiviral therapy
* Patients achieving sustained virologic response (SVR), defined as undetectable serum HCV RNA at week 12 off-therapy

Exclusion Criteria:

* Poor access to sites for venipuncture

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemodialysis patients who undergo antiviral therapy for hepatitis C virus infection and who achieve sustained virologic response
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Cumulative reinfection rate | Through study completion, an average of 3 years
  Time-dependent accumulative proportion of participants with evidence of resurgence of HCV viremia from the time point of viral clearance after antiviral therapy to the time point of last follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Hua Liu, MD, Principal Investigator — National Taiwan University Hospital
Locations (7):
- Taiwan (7):
  - National Taiwan University Hospital, Yun-Lin Branch, Douliu
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei City Hospital, Ren-Ai Branch, Taipei
  - Taipei Medical University Hospital, Taipei
  - Tri-Service General Hospital, Taipei